CLINICAL TRIAL: NCT01272544
Title: Oral Health of Individuals Who Attended a Mother-child Dental Care Program - Longitudinal Study
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Lucia de Fatima Almeida de Deus Moura, UFPI
Other Study IDs: mouraiso
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2009-09

CONDITIONS: Health Behavior
Keywords: Dental caries; Epidemiology; Gingivitis; Oral health
MeSH Terms: conditions — Health Behavior; Dental Caries; Gingivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- participation in a dental health program: Group 1 - children who participated to a dental health program Group 2 - children who did not participate to dental health program
- participation in a preventive program: Group 1 - children who participated to the preventive program Group 2 - children who did not participate

SUMMARY:
The aim of this longitudinal study was to assess the oral health of individuals attending a mother-child dental care program (PPPWB). The mean DMFT and GBI in the second phase and the control group were 0.75 and 6.75, 1.47 and 10.74, respectively. It was concluded that the individuals who attended the PPPWB had better oral health status than the control group. When the two phases of the study were compared, it was noted that the individuals in the second phase had better oral health, although they had a higher score for gingival bleeding.

DETAILED DESCRIPTION:
The aim of this longitudinal study was to assess the oral health of individuals attending a mother-child dental care program (PPPWB). Letters were sent to the 343 children who were examined in phase 1. One hundred and thirty nine individuals returned for the oral examination - experimental group (40.5%). The control group consisted of 139 individuals who did not receive dental care from the PPPWB. These individuals were paired to the experimental group according to their age and socio-demographic characteristics. Gingival bleeding (GBI) and DMFT indices were used in order to determine the children's oral health status. The mean DMFT and GBI in the second phase and the control group were 0.75 and 6.75, 1.47 and 10.74, respectively. It was concluded that the individuals who attended the PPPWB had better oral health status than the control group. When the two phases of the study were compared, it was noted that the individuals in the second phase had better oral health, although they had a higher score for gingival bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Children who participated to the program

Exclusion Criteria:

* children who did not participate

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Letters were sent to 343 of the examined children, inviting the guardians to take their children for an oral health assessment at the children's dental clinic at UFPI. The number of children that returned for an examination was 139, and these individuals comprised the experimental group.
  Control Group After assessing the characteristics of the experimental group, the control group was determined and consisted of 139 individuals (93 females and 46 males) who were paired to the experimental group according to their socio-demographic characteristics and age but who had not attended the PPPWB.
  The study hypothesis is that individuals who attended the PPPWB have better oral health than those who did not attend it.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2009-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucia D Moura, PhD, Study Chair — Universidade Federal do Piaui; Cacilda C Lima, DDS, Principal Investigator — Universidade Federal do Piaui; Marcoeli S Moura, PhD, Study Director — Universidade Federal do Piaui; Josilda F Martins, PhD, Study Director — Universidade Federal do Piaui; Marina M Lima, PhD, Study Director — Universidade Federal do Piaui